CLINICAL TRIAL: NCT06355583
Title: Intestinal Microbiota Transplant Prior to Allogeneic Stem Cell Transplant (MAST) Trial
Acronym: MAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C/42/2022; 2022-003617-10 (EudraCT Number)
Record Dates: First submitted 2023-10-03; First posted 2024-04-09 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Acute Lymphoblastic Leukaemia; Acute Leukemia of Ambiguous Lineage; Chronic Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Acute Myeloid Leukemia
Keywords: MAST
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Patients randomised on to the placebo arm will swallow 10 placebo capsules once at the second study visit approximately 2 weeks before the stem cell transplantation. The capsules contain inactive ingredients (microcrystalline cellulose and magnesium stearate) and will have the same appearance, weight, and packaging weight to the IMT capsules in the treatment arm to maintain treatment blinding.
  Interventions: Drug: Placebo
- EBX-102-02 (Active Comparator): Patients randomised on to the Treatment arm will swallow 10 capsules once at the second study visit approximately 2 weeks before the stem cell transplantation. Each capsule will contain 1x10^6 - 1x10^9 colony forming units (CFU)/g of viable microorganisms and will have the same appearance, weight and packaging weight to the placebo capsules in the treatment arm to maintain treatment blinding.
  Interventions: Drug: EBX-102

INTERVENTIONS:
Drug: EBX-102 — EBX-102 is a white size 0 gastro-resistant hydroxypropyl methylcellulose (HPMC) capsule containing communities of dried, intestinal microorganisms extracted from rigorously screened pooled human stool samples obtained from volunteer accredited donors.
  Other Names: IMT capsules
  Arms: EBX-102-02
Drug: Placebo — The capsules contain inactive ingredients microcrystalline cellulose and magnesium stearate.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test the ability to restore gut microbiota to healthier levels in patients with blood cancers scheduled to have stem cell transplant.

The main questions it aims to answer are:

* Tolerability and acceptability of intestinal microbiota transplantation (IMT) versus placebo (as assessed via patient perspective questionnaires
* Changes in gut microbiome diversity across all timepoints
* Markers of general health, infective/microbiological and haematological outcomes including, days of fever, admission to intensive care unit, survival, non-relapsed mortality, and incidence of graft-versus-host disease across all time points measured.

Participants will be asked at their routine follow up visits to,

* Provide stool, urine and blood samples at the scheduled study visits
* Complete questionnaires at selected visits
* Swallow either Placebo or IMT capsules once at the second study visit which will occur 2 weeks prior to the stem cell transplant (+/-3 days)

Researchers will compare IMT capsules and Placebo to investigate the change in gut microbiota diversity.

ELIGIBILITY:
Inclusion Criteria:

1. - Patients aged 18 years and over with a morphological documented diagnosis of ALL, acute myeloid leukemia (AML), AL of ambiguous lineage, myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), and CML in blast phase (Appendix 2) who are deemed fit for allogenic HCT with one of the following disease characteristics: ALL, AML, AL of ambiguous lineage

   * Patients in first complete remission (CR1) or second complete remission (CR2) including complete remission with incomplete blood count recovery with < 5% blasts (Appendix 2)
   * Secondary leukaemia (defined as previous history of MDS, antecedent haematological disease or chemotherapy exposure) in CR1 or CR2 defined as < 5% blasts (Appendix 2) MDS and CMML
   * Patients with advanced or high risk MDS with an International Prognostic Scoring System (IPSS-M) moderate high or higher including intermediate or high risk CMML who have < 5% blasts at the time of randomisation (Appendix 2) CML in blast phase
   * Patients with Philadelphia or BCR:ABL1 positive chronic myeloid leukaemia (CML) in blast phase defined by the presence of ≥ 20% blasts in blood or bone marrow who have achieved second chronic phase with < 5% blasts (Appendix 2).
2. Patients must have completed minimum of two cycles of intensive chemotherapy prior to trial enrolment (Appendix 1)
3. Patients must have received broad-spectrum antibiotics within 3 months prior to trial enrolment
4. Patients must be considered suitable/fit to undergo allogeneic hematopoietic cell transplantation (HCT) as clinically judged by the Local investigator
5. Patients with an Karnofsky performance status score 60 or above (Appendix 3)
6. Females of and male patients of reproductive potential (i.e., not post-menopausal or surgically sterilised) must use appropriate, highly effective, contraception from the point of commencing therapy until 6 months after treatment
7. Patients have given written informed consent
8. Patients willing and able to comply with scheduled study visits and laboratory tests

Exclusion Criteria:

1. Patients with contraindications to receiving allogeneic HCT.
2. Female patients who are pregnant or breastfeeding. All women of childbearing potential must have a negative pregnancy test before commencing treatment.
3. Adults of reproductive potential not willing to use appropriate, highly effective, contraception during the specified period.
4. Patients with renal or hepatic impairment as clinically judged by the Local Investigator.
5. Patients with active infection, HIV-positive or chronic active hepatitis B virus (HBV) or hepatitis C virus (HCV).
6. Patients with a concurrent active malignancy or a prior malignancy, except lobular breast carcinoma in situ, fully resected basal cell or squamous cell carcinoma of skin or treated cervical carcinoma in situ, incidental histologic finding of prostate cancer (T1a or T1b using the tumour, node, metastasis (TNM) clinical staging system), previous MDS, CMML, Myeloproliferative neoplasms (MPN) resulting in secondary AML. Cancer treated with curative intent ≥ 5 years previously will be allowed. Cancer treated with curative intent < 5 years previously will not be allowed.
7. Swallowing difficulties that may preclude safe use of IMT capsules.
8. Administration of IMT within 3 months prior to enrolment (probiotic administration prior to enrolment is allowed but should be recorded at screening).
9. Patients taking probiotics after enrolment to the trial.
10. Gastrointestinal disorders and diseases, including delayed gastric emptying, coeliac disease, cystic fibrosis, inflammatory bowel disease, irritable bowel syndrome, chronic diarrhoea, and colonic perforation or fistula.
11. Any autoimmune disease requiring, or that may require, systemic treatment with steroids and/or other immunosuppressants/immunomodulators.
12. Significant bleeding disorder (ALL, AML, AL of ambiguous lineage, MDS, CMML, and CML satisfying inclusion criteria are not excluded).
13. Anaphylactic food allergy.
14. Requirement for vasopressors.
15. Valvular heart disease or known structural defects of the heart.
16. Known severe allergy to capsule components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota diversity using Inverse Simpsons Index | Screening - up to 42 before stem cell transplantation (HCT) and Assessment 5 - Day 28(+/-3) post stem cell transplantation (HCT)
  Ecological metric to measure diversity in the gut microbiome in samples collected at two time points. It considers both the number of species present (richness) and their relative abundance (evenness). The Inverse index scale ranges from 0-1 with higher ranges indicating higher diversity.

SECONDARY OUTCOMES:
Gut Microbiome Diversity - Alpha diversity | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured via changes in Chao-1 , Shannon index and Faith's PD to estimate the richness and functional composition across all timepoints
Alpha Diversity - Chao1 Index | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  A non-parametric method for estimating Species Richness: referring to the total number of different species present in the gut microbiome, particularly useful for accounting for undetected species.points
Alpha Diversity - Shannon Index | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  An ecological metric used to measure which combines both, Species Richness: referring to the total number of different species present in the gut microbiome.
  Species Evenness: this indicates how evenly the species are distributed. A higher index value implies higher evenness and richness.
Alpha Diversity - Faiths Phylogenetic Diversity (Faiths PD) | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  An ecological metric used to measure, Species Richness: referring to the total number of different species present in the gut microbiome. Faiths PD also uses the phylogenetic tree of the identified species to measure the total evolutionary distance.
  A higher Faith's PD value indicates a wider range of evolutionary diversity
Beta Diversity - Aitchison Distance | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Ecological metric used to compare the distance in compositions in stool samples collected at different time points will with the baseline stool sample. Larger distances might indicate differences in bacterial communities present in the gut microbiome
Gut Microbiome Taxonomic Composition | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured using shallow shotgun sequencing which indicates the specific bacterial types and relative abundancies. stool samples collected at different time points will be compared with the baseline stool sample.
Markers of general health - ITU Admission | Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the total number days spent in an intensive care unit (ITU) from treatment to end of study
Quality of life EQ-5D-5L | Screening up to Day-42, Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Quality of live measured by standardised EQ-5D-5L questionnaire which assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression on a scale from 0 (worst health imaginable) to 100 (best health imaginable
Quality of Life EORTC-QLQ-C30 | Screening up to Day-42, Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Quality of life measured by standardised EORTC-QLQ-C3O Questionnaire Contains 30 questions grouped into 15 functional scales. Each scale is scored individually based on the answers, resulting in a score between 0 and 100. A higher score indicates better quality of life in that specific m
Infective Haematological Outcomes - Fever Occurrence | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Fever: Rise in body temperature above the normal range 38°C (100.4°F) or higher reported across all study time points post screening.
Infective Haematological Outcomes - Fever CTCAE Grade | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured by the number of reported occurrences of grade I - IV following the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grading system
Infective Haematological Outcomes - Infection | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured by reported occurrences of bloodstream infections and urinary tract infections across all time points.
Infective Haematological Outcomes - Multi drug Resistant Bacterial Colonisation (MDROs) | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the number of reported deaths not caused by relapse or progression
Infective Haematological Outcomes - Antibiotic Use | All timepoints, Screening up to Day-42, Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured by reported use of antibiotics to treat an infection diagnosis at all study timepoints.
Markers of General Health - Severity of Mucositis | The outcome will be assessed at Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the number of reported occurrences of mucositis grade III and above following the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) grading system post stem cell transplantation.
Markers of General Health -Occurrence of Severe Acute Kidney Injury (AKI) | The outcome will be assessed at Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the reported incidence of severe acute kidney post stem cell transplantation.
Markers of General Health - Occurrence of Severe liver dysfunction | The outcome will be assessed at Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the reported incidence of severe liver dysfunction post stem cell transplantation.
Markers of general health - Use of Parenteral Nutrition | The outcome will be assessed at Day -7(+/-2), Day 0(+/-1), Day 7(+/-3), Day 14(+/-3), Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured by the reported use of parenteral nutrition treatment post stem cell transplantation
Neutrophil and platelet engraftment data | Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Neutrophil and platelet engraftment data as defined by European Group for Blood and Marrow Transplantation (EBMT) will be routinely collected
Recovery of T-cell Chimaerisms, | Follow up Assessments: Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  T-cell count assessed by the lymphocyte subset analysis and immunoglobulin levels will be recorded at follow-up assessments.
Haematological Outcomes - Non-relapsed mortality | Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Assessed by the number of reported deaths not caused by relapse or progression post stem cell transplantation
Haematological Outcomes - Occurrence Graft vs Host Disease | Follow up Assessments: Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured by the reported occurrence of Graft vs Host Disease at all follow up assessments.
Haematological Outcomes - Severity of graft vs Host Disease | Follow up Assessments: Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Measured using the National Institutes of Health (NIH) Chronic/Acute GvHD Global Severity classification at all follow up assessments.
Overall Survival | Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Overall Survival (OS) - Measured from the time of the stem cell transplant date to the reporting of death from any cause up to 1 year post stem cell
Graft-versus disease-free relapse-free survival | Days Post HCT: Day 28(+/-3), Day 100(+/-7), Day 200(+/-7) & Day 365(+/-14)
  Graft-versus disease-free relapse-free survival (GFRS) - Measured from the time of the stem cell transplant date to the reporting of the first occurrence of either relapse or any grade of graft vs host disease (GVHD)

CONTACTS AND LOCATIONS:
Overall Officials: Jiri Pavlu, Principal Investigator — Imperial College London
Locations (8):
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Leeds Teaching Hospital NHS Trust, Leeds, England
  - University College London Hospitals NHS Trust, London, England
  - Kings College NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust, London, England
  - Royal Mardsen Hostpital, London
  - Manchester University NHS Foundation Trust, Manchester
  - Manchester University NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset may be prepared for sharing; a controlled access approach will be followed where data requestors will need to provide information to gain access to the data. The review will be taken by the sponsor and the clinical trials unit for a fully unbiased approach as recommended by the Institute of Medicine. Access to data may be granted but further restrictions regarding the access process may apply e.g. access through a secure web interface." The study protocol will be published as a supplement.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Study Protocol will be available once the study is open for recruitment Analytic code and Clinical Study Report can be requested once results have been published
Access Criteria: Data Requestors must contact the MAST study (mast-trial@imperial.ac.uk) to follow the approval process of obtaining access to the trial data

REFERENCES:
- [Background] Sargent DJ, Taylor JM. Current issues in oncology drug development, with a focus on Phase II trials. J Biopharm Stat. 2009;19(3):556-62. doi: 10.1080/10543400902802474. PMID 19384696
- [Background] Rubinstein LV, Korn EL, Freidlin B, Hunsberger S, Ivy SP, Smith MA. Design issues of randomized phase II trials and a proposal for phase II screening trials. J Clin Oncol. 2005 Oct 1;23(28):7199-206. doi: 10.1200/JCO.2005.01.149. PMID 16192604
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Malard F, Vekhoff A, Lapusan S, Isnard F, D'incan-Corda E, Rey J, Saillard C, Thomas X, Ducastelle-Lepretre S, Paubelle E, Larcher MV, Rocher C, Recher C, Tavitian S, Bertoli S, Michallet AS, Gilis L, Peterlin P, Chevallier P, Nguyen S, Plantamura E, Boucinha L, Gasc C, Michallet M, Dore J, Legrand O, Mohty M. Gut microbiota diversity after autologous fecal microbiota transfer in acute myeloid leukemia patients. Nat Commun. 2021 May 25;12(1):3084. doi: 10.1038/s41467-021-23376-6. PMID 34035290
- [Background] Taur Y, Coyte K, Schluter J, Robilotti E, Figueroa C, Gjonbalaj M, Littmann ER, Ling L, Miller L, Gyaltshen Y, Fontana E, Morjaria S, Gyurkocza B, Perales MA, Castro-Malaspina H, Tamari R, Ponce D, Koehne G, Barker J, Jakubowski A, Papadopoulos E, Dahi P, Sauter C, Shaffer B, Young JW, Peled J, Meagher RC, Jenq RR, van den Brink MRM, Giralt SA, Pamer EG, Xavier JB. Reconstitution of the gut microbiota of antibiotic-treated patients by autologous fecal microbiota transplant. Sci Transl Med. 2018 Sep 26;10(460):eaap9489. doi: 10.1126/scitranslmed.aap9489. PMID 30257956
- [Background] Peled JU, Gomes ALC, Devlin SM, Littmann ER, Taur Y, Sung AD, Weber D, Hashimoto D, Slingerland AE, Slingerland JB, Maloy M, Clurman AG, Stein-Thoeringer CK, Markey KA, Docampo MD, Burgos da Silva M, Khan N, Gessner A, Messina JA, Romero K, Lew MV, Bush A, Bohannon L, Brereton DG, Fontana E, Amoretti LA, Wright RJ, Armijo GK, Shono Y, Sanchez-Escamilla M, Castillo Flores N, Alarcon Tomas A, Lin RJ, Yanez San Segundo L, Shah GL, Cho C, Scordo M, Politikos I, Hayasaka K, Hasegawa Y, Gyurkocza B, Ponce DM, Barker JN, Perales MA, Giralt SA, Jenq RR, Teshima T, Chao NJ, Holler E, Xavier JB, Pamer EG, van den Brink MRM. Microbiota as Predictor of Mortality in Allogeneic Hematopoietic-Cell Transplantation. N Engl J Med. 2020 Feb 27;382(9):822-834. doi: 10.1056/NEJMoa1900623. PMID 32101664
- [Background] van Lier YF, Davids M, Haverkate NJE, de Groot PF, Donker ML, Meijer E, Heubel-Moenen FCJI, Nur E, Zeerleder SS, Nieuwdorp M, Blom B, Hazenberg MD. Donor fecal microbiota transplantation ameliorates intestinal graft-versus-host disease in allogeneic hematopoietic cell transplant recipients. Sci Transl Med. 2020 Aug 12;12(556):eaaz8926. doi: 10.1126/scitranslmed.aaz8926. PMID 32801142
- [Background] Shouval R, Geva M, Nagler A, Youngster I. Fecal Microbiota Transplantation for Treatment of Acute Graft-versus-Host Disease. Clin Hematol Int. 2019 Apr 18;1(1):28-35. doi: 10.2991/chi.d.190316.002. eCollection 2019 Mar. PMID 34595408
- [Background] DeFilipp Z, Peled JU, Li S, Mahabamunuge J, Dagher Z, Slingerland AE, Del Rio C, Valles B, Kempner ME, Smith M, Brown J, Dey BR, El-Jawahri A, McAfee SL, Spitzer TR, Ballen KK, Sung AD, Dalton TE, Messina JA, Dettmer K, Liebisch G, Oefner P, Taur Y, Pamer EG, Holler E, Mansour MK, van den Brink MRM, Hohmann E, Jenq RR, Chen YB. Third-party fecal microbiota transplantation following allo-HCT reconstitutes microbiome diversity. Blood Adv. 2018 Apr 10;2(7):745-753. doi: 10.1182/bloodadvances.2018017731. PMID 29592876
- [Background] Bloom PP, Luevano JM Jr, Miller KJ, Chung RT. Deep stool microbiome analysis in cirrhosis reveals an association between short-chain fatty acids and hepatic encephalopathy. Ann Hepatol. 2021 Nov-Dec;25:100333. doi: 10.1016/j.aohep.2021.100333. Epub 2021 Feb 20. PMID 33621653
- [Background] Staley C, Hamilton MJ, Vaughn BP, Graiziger CT, Newman KM, Kabage AJ, Sadowsky MJ, Khoruts A. Successful Resolution of Recurrent Clostridium difficile Infection using Freeze-Dried, Encapsulated Fecal Microbiota; Pragmatic Cohort Study. Am J Gastroenterol. 2017 Jun;112(6):940-947. doi: 10.1038/ajg.2017.6. Epub 2017 Feb 14. PMID 28195180
- [Background] Cammarota G, Ianiro G, Tilg H, Rajilic-Stojanovic M, Kump P, Satokari R, Sokol H, Arkkila P, Pintus C, Hart A, Segal J, Aloi M, Masucci L, Molinaro A, Scaldaferri F, Gasbarrini G, Lopez-Sanroman A, Link A, de Groot P, de Vos WM, Hogenauer C, Malfertheiner P, Mattila E, Milosavljevic T, Nieuwdorp M, Sanguinetti M, Simren M, Gasbarrini A; European FMT Working Group. European consensus conference on faecal microbiota transplantation in clinical practice. Gut. 2017 Apr;66(4):569-580. doi: 10.1136/gutjnl-2016-313017. Epub 2017 Jan 13. PMID 28087657
- [Background] Kao D, Roach B, Silva M, Beck P, Rioux K, Kaplan GG, Chang HJ, Coward S, Goodman KJ, Xu H, Madsen K, Mason A, Wong GK, Jovel J, Patterson J, Louie T. Effect of Oral Capsule- vs Colonoscopy-Delivered Fecal Microbiota Transplantation on Recurrent Clostridium difficile Infection: A Randomized Clinical Trial. JAMA. 2017 Nov 28;318(20):1985-1993. doi: 10.1001/jama.2017.17077. PMID 29183074
- [Background] Taur Y, Xavier JB, Lipuma L, Ubeda C, Goldberg J, Gobourne A, Lee YJ, Dubin KA, Socci ND, Viale A, Perales MA, Jenq RR, van den Brink MR, Pamer EG. Intestinal domination and the risk of bacteremia in patients undergoing allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2012 Oct;55(7):905-14. doi: 10.1093/cid/cis580. Epub 2012 Jun 20. PMID 22718773
- [Background] Innes AJ, Mullish BH, Ghani R, Szydlo RM, Apperley JF, Olavarria E, Palanicawandar R, Kanfer EJ, Milojkovic D, McDonald JAK, Brannigan ET, Thursz MR, Williams HRT, Davies FJ, Marchesi JR, Pavlu J. Fecal Microbiota Transplant Mitigates Adverse Outcomes Seen in Patients Colonized With Multidrug-Resistant Organisms Undergoing Allogeneic Hematopoietic Cell Transplantation. Front Cell Infect Microbiol. 2021 Aug 27;11:684659. doi: 10.3389/fcimb.2021.684659. eCollection 2021. PMID 34513724
- [Background] Mullish BH, Quraishi MN, Segal JP, McCune VL, Baxter M, Marsden GL, Moore DJ, Colville A, Bhala N, Iqbal TH, Settle C, Kontkowski G, Hart AL, Hawkey PM, Goldenberg SD, Williams HRT. The use of faecal microbiota transplant as treatment for recurrent or refractory Clostridium difficile infection and other potential indications: joint British Society of Gastroenterology (BSG) and Healthcare Infection Society (HIS) guidelines. Gut. 2018 Nov;67(11):1920-1941. doi: 10.1136/gutjnl-2018-316818. Epub 2018 Aug 28. PMID 30154172
- [Background] Shogbesan O, Poudel DR, Victor S, Jehangir A, Fadahunsi O, Shogbesan G, Donato A. A Systematic Review of the Efficacy and Safety of Fecal Microbiota Transplant for Clostridium difficile Infection in Immunocompromised Patients. Can J Gastroenterol Hepatol. 2018 Sep 2;2018:1394379. doi: 10.1155/2018/1394379. eCollection 2018. PMID 30246002
- [Background] Ghani R, Mullish BH, McDonald JAK, Ghazy A, Williams HRT, Brannigan ET, Mookerjee S, Satta G, Gilchrist M, Duncan N, Corbett R, Innes AJ, Pavlu J, Thursz MR, Davies F, Marchesi JR. Disease Prevention Not Decolonization: A Model for Fecal Microbiota Transplantation in Patients Colonized With Multidrug-resistant Organisms. Clin Infect Dis. 2021 Apr 26;72(8):1444-1447. doi: 10.1093/cid/ciaa948. PMID 32681643
- [Background] Woodhouse CA, Patel VC, Goldenberg S, Sanchez-Fueyo A, China L, O'Brien A, Flach C, Douiri A, Shawcross D. PROFIT, a PROspective, randomised placebo controlled feasibility trial of Faecal mIcrobiota Transplantation in cirrhosis: study protocol for a single-blinded trial. BMJ Open. 2019 Feb 15;9(2):e023518. doi: 10.1136/bmjopen-2018-023518. PMID 30772848
- [Background] Tan P, Li X, Shen J, Feng Q. Fecal Microbiota Transplantation for the Treatment of Inflammatory Bowel Disease: An Update. Front Pharmacol. 2020 Sep 18;11:574533. doi: 10.3389/fphar.2020.574533. eCollection 2020. PMID 33041818
- [Background] Tang Q, Jin G, Wang G, Liu T, Liu X, Wang B, Cao H. Current Sampling Methods for Gut Microbiota: A Call for More Precise Devices. Front Cell Infect Microbiol. 2020 Apr 9;10:151. doi: 10.3389/fcimb.2020.00151. eCollection 2020. PMID 32328469
- [Background] Hooper LV, Littman DR, Macpherson AJ. Interactions between the microbiota and the immune system. Science. 2012 Jun 8;336(6086):1268-73. doi: 10.1126/science.1223490. Epub 2012 Jun 6. PMID 22674334
- [Background] van der Waaij D, Berghuis JM, Lekkerkerk JE. Colonization resistance of the digestive tract of mice during systemic antibiotic treatment. J Hyg (Lond). 1972 Dec;70(4):605-10. doi: 10.1017/s0022172400022464. PMID 4567309
- [Background] Buffie CG, Bucci V, Stein RR, McKenney PT, Ling L, Gobourne A, No D, Liu H, Kinnebrew M, Viale A, Littmann E, van den Brink MR, Jenq RR, Taur Y, Sander C, Cross JR, Toussaint NC, Xavier JB, Pamer EG. Precision microbiome reconstitution restores bile acid mediated resistance to Clostridium difficile. Nature. 2015 Jan 8;517(7533):205-8. doi: 10.1038/nature13828. Epub 2014 Oct 22. PMID 25337874
- [Background] Hacquard S, Garrido-Oter R, Gonzalez A, Spaepen S, Ackermann G, Lebeis S, McHardy AC, Dangl JL, Knight R, Ley R, Schulze-Lefert P. Microbiota and Host Nutrition across Plant and Animal Kingdoms. Cell Host Microbe. 2015 May 13;17(5):603-16. doi: 10.1016/j.chom.2015.04.009. PMID 25974302
- [Background] Marchesi JR, Ravel J. The vocabulary of microbiome research: a proposal. Microbiome. 2015 Jul 30;3:31. doi: 10.1186/s40168-015-0094-5. eCollection 2015. PMID 26229597
- [Background] Human Microbiome Project Consortium. Structure, function and diversity of the healthy human microbiome. Nature. 2012 Jun 13;486(7402):207-14. doi: 10.1038/nature11234. PMID 22699609
- [Background] Eckburg PB, Bik EM, Bernstein CN, Purdom E, Dethlefsen L, Sargent M, Gill SR, Nelson KE, Relman DA. Diversity of the human intestinal microbial flora. Science. 2005 Jun 10;308(5728):1635-8. doi: 10.1126/science.1110591. Epub 2005 Apr 14. PMID 15831718
- [Derived] Mullish BH, Innes AJ, Roberts LA, Anim-Burton S, Webber L, Johnson NA, Ghani R, Farshi P, Khan AB, Kinsella F, Kottaridis P, Krishnamurthy P, Nicholson E, Palanicawandar R, Wheeler G, Davies F, Marchesi JR, Pavlu J. Intestinal Microbiota Transplant Prior to Allogeneic Stem Cell Transplant (MAST) trial: study protocol for a multicentre, double-blinded, placebo-controlled, phase IIa trial. BMJ Open. 2024 Dec 22;14(12):e093120. doi: 10.1136/bmjopen-2024-093120. PMID 39773995